CLINICAL TRIAL: NCT06500897
Title: Mid Term Follow up of VEST Device to Enhance Safein Vein Patency: a Multicentric Study
Brief Title: VEST Device to Enhance Safein Vein Patency
Status: Completed | Type: Observational
Sponsor: Cardiochirurgia E.H. (Other)
Responsible Party: Sponsor
Other Study IDs: EHMHVU-001
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Coronary Artery Bypass
Keywords: Coronary Artery Bypass; Safein Vein; Mesh support

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: VEST — External MEsh Support for safein vein

SUMMARY:
Purpose - Bypass grafting is the gold standard for severe coronary disease, yet most repeat revascularizations target previously grafted territories. External stenting of saphenous vein grafts, the most frequently used bypass conduit, has been shown to minimize disease markers. This study evaluates clinical outcomes of external stenting in real world routine practice.

Methods - Three centers enrolled a prospective real-world cohort of external- stenting- enhanced CABG patients. All patients received an internal mammary artery graft to the left anterior descending artery and additional arterial and/or venous grafts. One or more venous grafts were externally stented. Choice of conduits, use of cardiopulmonary bypass, and vein harvesting technique were performed according to the routine practice of each surgeon.

All patients were prescribed standard of care medication and were followed via on site visits or phone interviews for major adverse myocardial and cerebral effects.

ELIGIBILITY:
Inclusion Criteria:

* CABG with at least one VEST implant

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All comers for CABG with at least one vessel treated with VESTed Vein
Sampling Method: Non-Probability Sample
Enrollment: 385 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-08 (Actual)

PRIMARY OUTCOMES:
Re-rivascularization | Up to 7 years
  Number of PCI or re-CABG performed, stratified by target site
MACCE | Up to 7 years
  Major adverse cardiac and cerebrovascular events

CONTACTS AND LOCATIONS:
Overall Officials: Luca We, Principal Investigator — European Hospital - Rome
Locations (3):
- Medical University of Vienna, Vienna, Austria
- Italy (2):
  - Cardiochirurgia European Hospital, Rome
  - Mauriziano Hospital, Turin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sandner S, Angleitner P, Laufer G, Zimpfer D. External stent (VEST) for saphenous vein grafts in coronary artery bypass grafting. Multimed Man Cardiothorac Surg. 2019 Feb 1;2019. doi: 10.1510/mmcts.2019.007. PMID 30767438
- [Result] Weltert LP, Audisio K, Bellisaro A, Bardi G, Flocco R, De Paulis R, Centofanti P. External stenting of vein grafts in coronary artery bypass grating: interim results from a two centers prospective study. J Cardiothorac Surg. 2021 Apr 12;16(1):74. doi: 10.1186/s13019-021-01406-0. PMID 33845865
- [Result] Sandner SE, Donovan TJ, Edelstein S, Puskas JD, Angleitner P, Krasopoulos G, Channon K, Gehrig T, Rajakaruna C, Ladyshenskij L, De Silva R, Bonaros N, Bolotin G, Jacobs S, Thielmann M, Choi YH, Ohri S, Lipey A, Friedrich I, Taggart DP. Effects of the harvesting technique and external stenting on progression of vein graft disease 2 years after coronary artery bypass. Eur J Cardiothorac Surg. 2022 Jun 15;62(1):ezac045. doi: 10.1093/ejcts/ezac045. PMID 35312782